CLINICAL TRIAL: NCT05382325
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety and Tolerability of MK-1484 as a Monotherapy and in Combination With Pembrolizumab in Adult Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Study of MK-1484 as Monotherapy and in Combination With Pembrolizumab (MK-3475) In Advanced or Metastatic Solid Tumors (MK-1484-001)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1484-001; MK-1484-001 (Other: MSD); 2023-505067-36 (Registry Identifier: EU CT); 2021-005220-38 (EudraCT Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-1484 (Experimental): Participants will receive MK-1484 every 3 weeks (Q3W) or 21-day cycle at escalating dose levels from 0.2-60 mg for up to a total of 35 cycles (up to approximately 24 months).
  Interventions: Biological: MK-1484
- MK-1484 + Pembrolizumab (Experimental): Participants will receive MK-1484 Q3W at escalating dose levels from 10-60 mg plus pembrolizumab 200 mg once every 21-day cycle for up to a total of 35 cycles (up to approximately 24 months).
  Interventions: Biological: MK-1484; Biological: Pembrolizumab

INTERVENTIONS:
Biological: MK-1484 — Subcutaneous (SC) injection
  Other Names: SP'482
Biological: Pembrolizumab — Intravenous (IV) infusion
  Other Names: MK-3475; Keytruda®
  Arms: MK-1484 + Pembrolizumab

SUMMARY:
The purpose of this study is to assess the safety and tolerability and to establish a preliminary recommended Phase 2 dose (RP2D) of MK-1484 administered as monotherapy and in combination with pembrolizumab (MK-3475) in adults with advanced or metastatic solid tumors.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and has received, or been intolerant to, all treatment known to confer clinical benefit.
* Has measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by the local site investigator/radiology.
* Has normal cardiac function based on transthoracic echocardiogram (TTE) or multigated acquisition scan (MUGA)
* Has provided an evaluable archival or newly obtained tumor tissue sample for biomarker analysis.
* Has adequate organ function.
* A male participant must agree to use contraception and should refrain from donating sperm during the specified period(s) of at least 120 days after study interventions.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and at least 1 of the following: not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period for at least 120 days after study intervention.

Exclusion Criteria:

* Has and chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) before the first dose of study intervention, or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related AEs). Participants receiving ongoing replacement hormone therapy for endocrine immune-related AEs will not be excluded from participation in this study.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody and/or components of the study interventions.
* Has an active infection requiring therapy.
* Has a history of interstitial lung disease.
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy.
* Participants with known human immunodeficiency virus (HIV) and/or hepatitis B or C infections, or known to be positive for hepatitis B surface antigen (HBsAg)/hepatitis B virus (HBV) DNA or hepatitis C Antibody or ribonucleic acid (RNA).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, make administration of the study drugs hazardous, or make it difficult to monitor adverse effects such that it is not in the best interest of the participant to participate.
* Has known psychiatric or substance abuse disorders that would interfere with the participant's ability to cooperate with the requirements of the study.
* Has not fully recovered from any effects of major surgery without significant detectable infection. Surgeries that required general anesthesia must be completed at least 2 weeks before first study intervention administration. Surgery requiring regional/epidural anesthesia must be completed at least 72 hours before first study intervention administration and participants should be recovered.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the start of study treatment.
* Has had an allogeneic tissue/solid organ transplant in the last 5 years or has evidence of graft-versus-host disease.
* Has received any prior interleukin-2 (IL-2) based therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Dose-Limiting Toxicity (DLT) Graded Using National Cancer Institute Common Terminology Criteria for Adverse Events (AEs) Version 5.0 | Cycle 1 (Up to 21 days)
  DLT is defined as any of the following toxicities, if assessed by the investigator to be related to study treatment: Grade (Gr) 4 nonhematologic toxicity (not laboratory); Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia: Gr 4 thrombocytopenia of any duration; Gr 3 thrombocytopenia associated with clinically significant bleeding; Gr 4 anemia regardless of duration; Nonhematologic AE Gr ≥3 in severity, with exceptions; Any Gr 3 or 4 nonhematologic laboratory abnormality if: clinically significant medical intervention is required, or if abnormality leads to hospitalization, persists for >1 week or results in drug-induced liver injury with exceptions; Gr 3 or Gr 4 febrile neutropenia; Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity; Treatment-related toxicity resulting in participant study treatment discontinuation during Cycle 1; Missing >25% of the MK-1484 dose during Cycle 1 resulting from treatment-related AE; Gr 5 toxicity.
Number of Participants Who Experience At Least One AE | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of MK-1484 | At designated time points (Up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine AUC.
Minimum Serum Concentration (Cmin) of MK-1484 | At designated time points (Up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmin.
Maximum Serum Concentration (Cmax) of MK-1484 | At designated time points (Up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- United States (2):
  - Sanford Cancer Center ( Site 0005), Sioux Falls, South Dakota
  - NEXT Oncology ( Site 0001), San Antonio, Texas
- Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0011), Toronto, Ontario, Canada
- Israel (2):
  - Rambam Health Care Campus-Oncology ( Site 0021), Haifa
  - Sheba Medical Center-ONCOLOGY ( Site 0020), Ramat Gan
- Netherlands (3):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 0035), Amsterdam, North Holland
  - Erasmus Medisch Centrum-Medical Oncology ( Site 0036), Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 0037), Utrecht

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26211&tenant=MT_MSD_9011